CLINICAL TRIAL: NCT05083104
Title: Assessment of the Natural Anticoagulant Profile in Patients With COVID-19
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Alaa Yousry Rageh, Resident of clinical and Chemical pathology, Sohag University
Other Study IDs: Soh-Med-21-10-09
Record Dates: First submitted 2021-10-13; First posted 2021-10-19 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: COVID-19 Patients

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- age and sex matched healthy control individuals.: controls divided into groups ,each group match in age and sex with cases
  Interventions: Diagnostic Test: laboratory investigations on coagulation profiles
- mild and severe cases of COVID 19 patients: Covid 19 cases diagnosed by PCR , mild cases have symptoms as fever, dry cough, and diarrhea and severe cases admitted in ICU
  Interventions: Diagnostic Test: laboratory investigations on coagulation profiles

INTERVENTIONS:
Diagnostic Test: laboratory investigations on coagulation profiles — CBC ,PT ,aPTT ,Protein C .Protein S ,ATIII and vWF

SUMMARY:
At the beginning of 2020, coronavirus disease 19 (COVID-19) was declared a pandemic of international concern and an unprecedented challenge for country-specific health care systems . Patients infected with COVID-19 develop from mild, self-limiting respiratory tract illness to severe progressive pneumonia associated with multi-organ failure . In particular, COVID-19 has been shown to exert significant effects on the hematopoietic system and hemostasis

DETAILED DESCRIPTION:
At the beginning of 2020, coronavirus disease 19 (COVID-19) was declared a pandemic of international concern and an unprecedented challenge for country-specific health care systems. The clinical feature of the disease is very wide and ranges from minor unspecified symptoms (such as fever, dry cough, and diarrhea) to severe pneumonia, lung insufficiency, and death. Fall in respiratory insufficiency needing mechanical ventilation, or in multiple organ failure occurs in 5% of the infected patients, mainly according to age and comorbidities. Coronaviruses are important pathogens in humans that can cause diseases ranging from the common cold to more severe and even fatal respiratory infections. Since the outbreak of the novel COVID-19 caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) in December 2019 in Wuhan, China, more than 2 million cases have been diagnosed globally to date and the number is still growing rapidly . Patients infected with COVID-19 develop from mild, self-limiting respiratory tract illness to severe progressive pneumonia associated with multi-organ failure .

Most of the people who contracted COVID-19 presented with mild symptoms (80.9%), then severe (13.8%), and finally critical (4.7%). Most of the confirmed cases were between the ages of 30 and 70 (86.6%), diagnosed in Hubei (74.7%), with an overall fatality rate of 2.3%, and 0.3% in health workers. The case fatality rate for critical cases was 49.0%. Patients with underlying diseases had much higher fatality rates than patients with no underlying diseases (10.5% for cardiovascular disease, 7.3% for diabetes, 6.3% for chronic respiratory disease, 6.0% for hypertension, 5.6% for cancer, and 0.9% for none).

In clinical practice, coagulation dysfunction is commonly found in COVID-19 patients, and the symptoms range from mild disorders of coagulation indicators to disseminated intravascular coagulation (DIC). The exact etiology of COVID-19-associated coagulopathy is unclear, diverse and multifactorial, and may include direct attack by the SARS-CoV-2 on vascular endothelial cells, cytokine storm-mediated inflammation-coagulation cascades, hypoxia, and complication with sepsis. Coagulation dysfunction or thrombocytopenia is closely associated with the severity and poor prognosis in COVID-19 patients .

Recently, coagulopathy was reported widely present in severe SARS-CoV-2 infected patients, and disseminated intravascular coagulation (DIC) developed in the majority of non-survivors . In particular, COVID-19 has been shown to exert significant effects on the hematopoietic system and hemostasis . Studies have emphasized that patients diagnosed with COVID-19 are susceptible to hypercoagulation and thrombotic events. Microvascular thrombosis has been observed in autopsies performed on patients .

Recent observations suggest that respiratory failure in coronavirus disease 2019 (COVID 19) infections are not caused by the development of the acute respiratory distress syndrome (ARDS) alone, but that microvascular thrombotic processes may contribute, also. One of the most significant poor prognostic signs in those patients is the development of coagulopathy .

ELIGIBILITY:
Inclusion Criteria:

* This study will be conducted on a group of patients who are diagnosed as COVID-19 by PCR, a group of them have mild symptoms and another group admitted in ICU (critically ill patients).

Exclusion Criteria:

* Any clinical condition cause hypercoagulability state such as:

  * Pregnancy.
  * Recent trauma or surgery.
  * Prolonged bed rest or immobility.
  * Cancer or its medications, such as tamoxifen, bevacizumab, thalidomide and lenalidomide.
  * Hormone replacement therapy.
  * Heparin-induced thrombocytopenia (decreased platelets in the blood due to heparin or low molecular weight heparin preparations).
  * Previous history of deep vein thrombosis or pulmonary embolism.
  * Myeloproliferative disorders such as polycythemia vera or essential thrombocytosis.

Ages: 5 Years to 50 Years | Sex: All
Age Groups: Child, Adult
Study Population: Group (I): represents the healthy control individuals Group (II): represents the mild and severe cases of COVID 19 patients.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Assess the effect of COVID-19 disease on coagulation cascade in patients of this disease. | within the same day of collection of samples
  The study will be conducted on a group of patients who are diagnosed as COVID-19 by PCR, All patients and controls were subjected to Full history taking ,clinical examination
Assess the effect of COVID-19 disease on coagulation cascade in patients of this disease. | within the same day of collection of samples
  The study will be conducted on a group of patients who are diagnosed as COVID-19 by PCR, and All patients and controls were subjected to Laboratory investigations as Complete blood count with platelet indices (MPV measured by fL & PDW measured by fL) ,
Assess the effect of COVID-19 disease on coagulation cascade in patients of this disease. | within the same day of collection of samples
  The study will be conducted on a group of patients who are diagnosed as COVID-19 by PCR, and All patients and controls were subjected to Laboratory investigations as Prothrombin time PT measured by seconds and activated partial thromboplastin time aPTT measured by seconds
Assess the effect of COVID-19 disease on coagulation cascade in patients of this disease. | within the same day of collection of samples
  The study will be conducted on a group of patients who are diagnosed as COVID-19 by PCR, and All patients and controls were subjected to Laboratory investigations as Protein C measured by %, Protein S measured by %, and Antithrombin III measured by %.
Assess the effect of COVID-19 disease on coagulation cascade in patients of this disease. | within the same day of collection of samples
  The study will be conducted on a group of patients who are diagnosed as COVID-19 by PCR, and All patients and controls were subjected to Laboratory investigations as von Willebrand factor vWF measured by IU per dL.